CLINICAL TRIAL: NCT02851953
Title: Effectiveness and Safety Evaluation of Aqueduct -100 Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqueduct Medical Ltd (Industry)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQD 01-15
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Cervix Uteri Dilation
Keywords: cervix, cervical dilation, balloon catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aqueduct 100 dilation (Experimental): Uterine cervix dilation through Aqueduct-100 device
  Interventions: Device: Aqueduct-100

INTERVENTIONS:
Device: Aqueduct-100

SUMMARY:
The purpose of the present clinical investigation is to collect data regarding the safety and effectiveness of the Aqueduct 100 device.

The effectiveness of the Aqueduct 100 will be determined by evaluating the ability to reach desired cervical dilation, and the time frame required to reach desired cervical dilation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, females, 18 years of age or older.
2. Subjects undergoing any process that requires dilation (intrauterine procedures).
3. Subjects understanding the nature of the study and willing to sign informed consent form.

Exclusion Criteria:

1. Subjects younger than 18 years of age.
2. Subject with the following infectious diseases: HIV, HBV, HCV, Syphilis.
3. Subject has been treated with any cervix dilating agent within 2 months before the screening.
4. Known contraindications or hypersensitivity to the components of the investigational product.
5. The patient has a condition or a concurrent severe and/or uncontrolled medical disease which could compromise participation, compliance with, and/or completion with study procedures.
6. Subjects undergoing abortion <7 and >9 weeks of pregnancy.
7. Subjects unwilling to sign the informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with dilation of cervix to a pre-determined diameter before the intrauterine procedure using Aqueduct-100 device. | Through study completion, approximately 9 months
  The primary outcome of this study is to determine the effectiveness of the Aqueduct-100 device to dilate the uterine cervices to the desired diameter.

SECONDARY OUTCOMES:
Occurrence of Adverse Events: rate, list and severity of AEs and SAEs. | Through study completion, approximately 9 months
  In vivo safety evaluation of using Aqueduct-100.
Time frame required to reach desired cervical dilation from start time (insertion of device) to completion of dilation (removal of catheter) | Through study completion, approximately 9 months
  Duration of the dilation procedure.
Measurement of physicians' satisfaction with the device, through the use of a questionnaire. | Through study completion, approximately 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Venturini, Professor, Principal Investigator — IRCCS AZIENDA OSPEDALIERA UNIVERSITARIA SAN MARTINO IST; Simone Ferrero, Professor, Study Director — IRCCS AZIENDA OSPEDALIERA UNIVERSITARIA SAN MARTINO IST
Locations (1):
- Irccs Azienda Ospedaliera Universitaria San Martino Ist, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazza E, Nava A, Bauer M, Winter R, Bajka M, Holzapfel GA. Mechanical properties of the human uterine cervix: an in vivo study. Med Image Anal. 2006 Apr;10(2):125-36. doi: 10.1016/j.media.2005.06.001. Epub 2005 Sep 6. PMID 16143559
- [Background] Buhimschi, C.; Buhimschi, I.; Malinow, A.; Saade, G.; Garfield, R.; Weiner, C., The Forces of Labour. Fetal and Maternal Medicine Review 2003, 14 (4), 273-307.
- [Background] Myers KM, Paskaleva AP, House M, Socrate S. Mechanical and biochemical properties of human cervical tissue. Acta Biomater. 2008 Jan;4(1):104-16. doi: 10.1016/j.actbio.2007.04.009. Epub 2007 Sep 27. PMID 17904431
- [Background] Kenyon NJ, Stevens JC, Stewart P, Black MM, Clifford A. A critical investigation of the measurement of the force required to dilate the human uterine cervix. Clin Phys Physiol Meas. 1988 May;9(2):155-61. doi: 10.1088/0143-0815/9/2/008. PMID 3391017
- [Background] S. Febvay, S. Socrate and M.D. House. Biomechanical modeling of cervical tissue. A quantitative investigation of cervical funneling. Proceedings of the ASME 2003 International Mechanical Engineering Congress and Exposition, Washington, D.C., November 2003.
- [Background] Arsenijevic S, Vukcevic-Globarevic G, Volarevic V, Macuzic I, Todorovic P, Tanaskovic I, Mijailovic M, Raicevic S, Jeremic B. Continuous controllable balloon dilation: a novel approach for cervix dilation. Trials. 2012 Oct 22;13:196. doi: 10.1186/1745-6215-13-196. PMID 23088906
- [Background] Nicolaides KH, Welch CC, MacPherson MB, Johnson IR, Filshie GM. Lamicel: a new technique for cervical dilatation before first trimester abortion. Br J Obstet Gynaecol. 1983 May;90(5):475-9. doi: 10.1111/j.1471-0528.1983.tb08947.x. PMID 6849849